CLINICAL TRIAL: NCT01059006
Title: Peripheral PresbyLASIK Using the Allegretto Wavelight System For The Treatment of Presbyopia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lead researcher completed fellowship and never got study off ground
Sponsor: University of California, San Diego (Other)
Responsible Party: David Schanzlin, MD, UCSD Shiley Eye Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 091460
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Refractive Error; Presbyopia
Keywords: Reflective Surgery; Presbyopia; PresbyLASIK
MeSH Terms: conditions — Refractive Errors; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PresbyLASIK (Experimental): Male or female patients with presbyopic symptoms who underwent PresbyLASIK.
  Interventions: Procedure: PresbyLASIK

INTERVENTIONS:
Procedure: PresbyLASIK — PresbyLASIK essentially involves the creation of a multifocal surface able to correct any visual defect for distance while simultaneously allowing freedom from near spectacle dependency in presbyopic patients.
  Other Names: Presbyopia; Presbyopic Symptoms

SUMMARY:
The aim of this study is to analyze the results of PresbyLASIK performed using the wavefront-optimized LASIK for the treatment of presbyopia on low hyperopic and low myopic patients with astigmatism. Visual performance will be assessed using clinical outcome measures of the following: refraction, near, intermediate and distance visual acuity, stereoacuity and contrast sensitivity. Questionnaires will also be used to evaluate how the patient's vision is before and after surgery.

DETAILED DESCRIPTION:
Presbyopia is a physiologic change related to age in which there is reduction in the eye's ability to focus in order to obtain clear vision for near distance. At approximately age 40 the range of accommodation begins to decrease and there is a diminishing capacity of the eye to focus on the nearest point it can focus on. This makes the need for corrective lenses a necessity in order to read at near as well as focus at an intermediate distance.

Presbyopia correction is one of the most frequently discussed topics in refractive surgery today. The idea of a creating a multifocal cornea using refractive surgery has sparked tremendous interest in finding a solution for this growing population throughout the world, especially amongst surgeons and the ophthalmic industry

PresbyLASIK essentially involves the creation of a multifocal surface able to correct any visual defect for distance while simultaneously allowing freedom from near spectacle dependency in presbyopic patients. PresbyLASIK is currently being offered routinely to patients in the San Diego area, across the country as well as in numerous centers around the world.

Conclusions from this study would serve as a guide for keratorefractive surgeons, who are pursuing peripheral PresbyLASIK, in determining the preoperative patient features in order to achieve the best outcome using the Wavelight-Allegretto System.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any race, and at least 35 to 80 years old with significant presbyopic symptoms at the time of the preoperative examination, and have signed an informed consent. The lower age limit of 35 is the earliest age in which reduction in accommodation occurs.
* Refractive error between +3.00 to -5.00 diopters (D) sphere at the spectacle plane with no more than 3.00D of refractive astigmatism (negative cylinder format)
* Best spectacle corrected visual acuity of at least 20/20 and J3 in both eyes.
* Residual corneal bed thickness of ≥ to 330 microns
* Demonstrated refractive stability, confirmed by clinical records. Neither the spherical nor the cylindrical portion of the refraction may have changed more than 0.50D during the 12-month period immediately preceding the baseline examination.
* Soft contact lens users must have removed their lenses at least one week before baseline measurements. Hard contact lens users (PMMA or rigid gas permeable lenses) must have removed their lenses at least 4 weeks prior to baseline measurements and have two central keratometry readings and two manifest refractions taken at least one week apart that do not differ by more than 0.50 diopter in either meridian; mires should be regular.
* Located in the greater San Diego area for a 6-month period.
* Exhibit strong motivation for attending the follow-up visits.
* Access to transportation to meet follow-up requirements.

Exclusion Criteria:

* Patients that have previously been treated for refractive surgery (LASIK and/or PRK)
* Patients with known history or have concurrent dry eye disease (e.g. keratoconjunctivitis sicca)
* Patients who have less than 5 mm pupil size in dimlight
* Female subjects who are pregnant, breast-feeding or intend to become pregnant during the first six months of the study.
* Concurrent topical or systemic medications that may impair healing, including corticosteroids, antimetabolites, isotretinoin (Accutane), amiodarone hydrochloride (Cordarone) and/or sumatriptan (Imitrex) or any other triptan.
* Medical condition(s), which, in the judgment of the investigator, may impair healing, including but not limited to: collagen vascular disease, autoimmune disease, immunodeficiency diseases, and ocular herpes zoster or simplex.
* Active ophthalmic disease, neovascularization of the cornea within 1mm of the intended ablation zone, or lens opacity.
* Evidence of glaucoma or an intraocular pressure greater than 22 mm Hg at baseline.
* Evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye.
* Corneal thickness insufficient to allow the residual remaining stromal bed to be at least 300 microns in each eye. The residual stromal bed thickness will be determined by subtracting both the LASIK flap thickness and depth of the ablation from the total central corneal thickness measured by pachymetry

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Uncorrected near visual acuity | 1 Day, 1 Week, 3 and 6 Months
Best corrected near visual acuity | 1 Day, 1 Week, 3 and 6 Months
Intermediate visual acuity | 1 Day, 1 Week, 3 and 6 Months
Stereoacuity test | 1 Day, 1 Week, 3 and 6 Months
Psychometric questionnaire | 1 Day, 1 Week, 3 and 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: David J Schanzlin, MD, Principal Investigator — UCSD Shiley Eye Center

REFERENCES:
- [Background] Epstein RL, Gurgos MA. Presbyopia treatment by monocular peripheral presbyLASIK. J Refract Surg. 2009 Jun;25(6):516-23. doi: 10.3928/1081597X-20090512-05. PMID 19603619
- [Background] Alio JL, Amparo F, Ortiz D, Moreno L. Corneal multifocality with excimer laser for presbyopia correction. Curr Opin Ophthalmol. 2009 Jul;20(4):264-71. doi: 10.1097/icu.0b013e32832a7ded. PMID 19537363
- [Background] Pinelli R, Ortiz D, Simonetto A, Bacchi C, Sala E, Alio JL. Correction of presbyopia in hyperopia with a center-distance, paracentral-near technique using the Technolas 217z platform. J Refract Surg. 2008 May;24(5):494-500. doi: 10.3928/1081597X-20080501-07. PMID 18494342
- [Background] Illueca C, Alio JL, Mas D, Ortiz D, Perez J, Espinosa J, Esperanza S. Pseudoaccommodation and visual acuity with Technovision presbyLASIK and a theoretical simulated Array multifocal intraocular lens. J Refract Surg. 2008 Apr;24(4):344-9. doi: 10.3928/1081597X-20080401-05. PMID 18500082
- [Background] Ortiz D, Alio JL, Illueca C, Mas D, Sala E, Perez J, Espinosa J. Optical analysis of presbyLASIK treatment by a light propagation algorithm. J Refract Surg. 2007 Jan;23(1):39-44. doi: 10.3928/1081-597X-20070101-07. PMID 17269242
- [Background] Alio JL, Chaubard JJ, Caliz A, Sala E, Patel S. Correction of presbyopia by technovision central multifocal LASIK (presbyLASIK). J Refract Surg. 2006 May;22(5):453-60. doi: 10.3928/1081-597X-20060501-06. PMID 16722483